CLINICAL TRIAL: NCT00535743
Title: A Multi-Center, Randomized, Safety Assessor-Blinded, Placebo- Controlled, Phase II, Parallel Dose-Finding Trial in Subjects of ASA 1-3 to Assess the Efficacy and Safety of 5 Doses of Sugammadex Administered at 3 and 15 Minutes After Administration of 1.0 and 1.2 mg/kg Rocuronium Bromide
Brief Title: Dose-Finding Trial With Sugammadex Administered at 3 and 15 Minutes After 1.0 and 1.2 mg/kg Rocuronium Bromide in Participants of ASA Class 1-3 (P05944; MK-8616-024)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P05944; 19.4.206 (Other: Organon Protocol Number); MK-8616-024 (Other: Merck Protocol Number)
Record Dates: First submitted 2007-09-25; First posted 2007-09-26 (Estimated); Results first posted 2019-02-11 (Actual); Last update posted 2019-02-11 (Actual); Status verified 2018-09

CONDITIONS: Anesthesia, General
MeSH Terms: interventions — Sugammadex; Sodium Chloride; Rocuronium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (24):
- Arm A. Placebo; 3 min after 1 mg/kg Esmeron® (Placebo Comparator): Placebo (single intravenous (IV) bolus) administered 3 minutes (min) after the bolus intubation dose of 1 mg/kg Esmeron®.
  Interventions: Drug: Placebo; Drug: Esmeron®
- Arm B. 2 mg/kg sugammadex; 3 min after 1 mg/kg Esmeron® (Experimental): Sugammadex (2 mg/kg; single IV bolus) administered 3 min after the bolus intubation dose of 1 mg/kg Esmeron®.
  Interventions: Drug: Sugammadex; Drug: Esmeron®
- Arm C. 4 mg/kg sugammadex; 3 min after 1 mg/kg Esmeron® (Experimental): Sugammadex (4 mg/kg; single IV bolus) administered 3 min after the bolus intubation dose of 1 mg/kg Esmeron®.
  Interventions: Drug: Sugammadex; Drug: Esmeron®
- Arm D. 8 mg/kg sugammadex; 3 min after 1 mg/kg Esmeron® (Experimental): Sugammadex (8 mg/kg; single IV bolus) administered 3 min after the bolus intubation dose of 1 mg/kg Esmeron®.
  Interventions: Drug: Sugammadex; Drug: Esmeron®
- Arm E. 12 mg/kg sugammadex; 3 min after 1 mg/kg Esmeron® (Experimental): Sugammadex (12 mg/kg; single IV bolus) administered 3 min after the bolus intubation dose of 1 mg/kg Esmeron®.
  Interventions: Drug: Sugammadex; Drug: Esmeron®
- Arm F. 16 mg/kg sugammadex; 3 min after 1 mg/kg Esmeron® (Experimental): Sugammadex (16 mg/kg; single IV bolus) administered 3 min after the bolus intubation dose of 1 mg/kg Esmeron®.
  Interventions: Drug: Sugammadex; Drug: Esmeron®
- Arm G. Placebo; 15 min after 1 mg/kg Esmeron® (Placebo Comparator): Placebo (single intravenous (IV) bolus) administered 15 min after the bolus intubation dose of 1 mg/kg Esmeron®.
  Interventions: Drug: Placebo; Drug: Esmeron®
- Arm H. 2 mg/kg sugammadex; 15 min after 1 mg/kg Esmeron® (Experimental): Sugammadex (2 mg/kg; single IV bolus) administered 15 min after the bolus intubation dose of 1 mg/kg Esmeron®.
  Interventions: Drug: Sugammadex; Drug: Esmeron®
- Arm I. 4 mg/kg sugammadex; 15 min after 1 mg/kg Esmeron® (Experimental): Sugammadex (4 mg/kg; single IV bolus) administered 15 min after the bolus intubation dose of 1 mg/kg Esmeron®.
  Interventions: Drug: Sugammadex; Drug: Esmeron®
- Arm J. 8 mg/kg sugammadex; 15 min after 1 mg/kg Esmeron® (Experimental): Sugammadex (8 mg/kg; single IV bolus) administered 15 min after the bolus intubation dose of 1 mg/kg Esmeron®.
  Interventions: Drug: Sugammadex; Drug: Esmeron®
- Arm K. 12 mg/kg sugammadex; 15 min after 1 mg/kg Esmeron® (Experimental): Sugammadex (12 mg/kg; single IV bolus) administered 15 min after the bolus intubation dose of 1 mg/kg Esmeron®.
  Interventions: Drug: Sugammadex; Drug: Esmeron®
- Arm L. 16 mg/kg sugammadex; 15 min after 1 mg/kg Esmeron® (Experimental): Sugammadex (16 mg/kg; single IV bolus) administered 15 min after the bolus intubation dose of 1 mg/kg Esmeron®.
  Interventions: Drug: Sugammadex; Drug: Esmeron®
- Arm M. Placebo; 3 min after 1.2 mg/kg Esmeron® (Placebo Comparator): Placebo (single IV bolus) administered 3 min after the bolus intubation dose of 1.2 mg/kg Esmeron®.
  Interventions: Drug: Placebo; Drug: Esmeron®
- Arm N. 2 mg/kg sugammadex; 3 min after 1.2 mg/kg Esmeron® (Experimental): Sugammadex (2 mg/kg; single IV bolus) administered 3 min after the bolus intubation dose of 1.2 mg/kg Esmeron®.
  Interventions: Drug: Sugammadex; Drug: Esmeron®
- Arm O. 4 mg/kg sugammadex; 3 min after 1.2 mg/kg Esmeron® (Experimental): Sugammadex (4 mg/kg; single IV bolus) administered 3 min after the bolus intubation dose of 1.2 mg/kg Esmeron®.
  Interventions: Drug: Sugammadex; Drug: Esmeron®
- Arm P. 8 mg/kg sugammadex; 3 min after 1.2 mg/kg Esmeron® (Experimental): Sugammadex (8 mg/kg; single IV bolus) administered 3 min after the bolus intubation dose of 1.2 mg/kg Esmeron®.
  Interventions: Drug: Sugammadex; Drug: Esmeron®
- Arm Q. 12 mg/kg sugammadex; 3 min after 1.2 mg/kg Esmeron® (Experimental): Sugammadex (12 mg/kg; single IV bolus) administered 3 min after the bolus intubation dose of 1.2 mg/kg Esmeron®.
  Interventions: Drug: Sugammadex; Drug: Esmeron®
- Arm R. 16 mg/kg sugammadex; 3 min after 1.2 mg/kg Esmeron® (Experimental): Sugammadex (16 mg/kg; single IV bolus) administered 3 min after the bolus intubation dose of 1.2 mg/kg Esmeron®.
  Interventions: Drug: Sugammadex; Drug: Esmeron®
- Arm S. Placebo; 15 min after 1.2 mg/kg Esmeron® (Placebo Comparator): Placebo (single IV bolus) administered 15 min after the bolus intubation dose of 1.2 mg/kg Esmeron®.
  Interventions: Drug: Placebo; Drug: Esmeron®
- Arm T. 2 mg/kg sugammadex; 15 min after 1.2 mg/kg Esmeron® (Experimental): Sugammadex (2 mg/kg; single IV bolus) administered 15 min after the bolus intubation dose of 1.2 mg/kg Esmeron®.
  Interventions: Drug: Sugammadex; Drug: Esmeron®
- Arm U. 4 mg/kg sugammadex; 15 min after 1.2 mg/kg Esmeron® (Experimental): Sugammadex (4 mg/kg; single IV bolus) administered 15 min after the bolus intubation dose of 1.2 mg/kg Esmeron®.
  Interventions: Drug: Sugammadex; Drug: Esmeron®
- Arm V. 8 mg/kg sugammadex; 15 min after 1.2 mg/kg Esmeron® (Experimental): Sugammadex (8 mg/kg; single IV bolus) administered 15 min after the bolus intubation dose of 1.2 mg/kg Esmeron®.
  Interventions: Drug: Sugammadex; Drug: Esmeron®
- Arm W. 12 mg/kg sugammadex; 15 min after 1.2 mg/kg Esmeron® (Experimental): Sugammadex (12 mg/kg; single IV bolus) administered 15 min after the bolus intubation dose of 1.2 mg/kg Esmeron®.
  Interventions: Drug: Sugammadex; Drug: Esmeron®
- Arm X. 16 mg/kg sugammadex; 15 min after 1.2 mg/kg Esmeron® (Experimental): Sugammadex (16 mg/kg; single IV bolus) administered 15 min after the bolus intubation dose of 1.2 mg/kg Esmeron®.
  Interventions: Drug: Sugammadex; Drug: Esmeron®

INTERVENTIONS:
Drug: Sugammadex — Sugammadex administered as a fast IV bolus dose (within 30 seconds) at 3 or 15 minutes following administration of Esmeron®, dosed at 2, 4, 8, 12 or 16 mg/kg according to participant actual body weight.
  Other Names: Org 25969; MK-8616; BRIDION®
  Arms: Arm B. 2 mg/kg sugammadex; 3 min after 1 mg/kg Esmeron®; Arm C. 4 mg/kg sugammadex; 3 min after 1 mg/kg Esmeron®; Arm D. 8 mg/kg sugammadex; 3 min after 1 mg/kg Esmeron®; Arm E. 12 mg/kg sugammadex; 3 min after 1 mg/kg Esmeron®; Arm F. 16 mg/kg sugammadex; 3 min after 1 mg/kg Esmeron®; Arm H. 2 mg/kg sugammadex; 15 min after 1 mg/kg Esmeron®; Arm I. 4 mg/kg sugammadex; 15 min after 1 mg/kg Esmeron®; Arm J. 8 mg/kg sugammadex; 15 min after 1 mg/kg Esmeron®; Arm K. 12 mg/kg sugammadex; 15 min after 1 mg/kg Esmeron®; Arm L. 16 mg/kg sugammadex; 15 min after 1 mg/kg Esmeron®; Arm N. 2 mg/kg sugammadex; 3 min after 1.2 mg/kg Esmeron®; Arm O. 4 mg/kg sugammadex; 3 min after 1.2 mg/kg Esmeron®; Arm P. 8 mg/kg sugammadex; 3 min after 1.2 mg/kg Esmeron®; Arm Q. 12 mg/kg sugammadex; 3 min after 1.2 mg/kg Esmeron®; Arm R. 16 mg/kg sugammadex; 3 min after 1.2 mg/kg Esmeron®; Arm T. 2 mg/kg sugammadex; 15 min after 1.2 mg/kg Esmeron®; Arm U. 4 mg/kg sugammadex; 15 min after 1.2 mg/kg Esmeron®; Arm V. 8 mg/kg sugammadex; 15 min after 1.2 mg/kg Esmeron®; Arm W. 12 mg/kg sugammadex; 15 min after 1.2 mg/kg Esmeron®; Arm X. 16 mg/kg sugammadex; 15 min after 1.2 mg/kg Esmeron®
Drug: Placebo — 0.9% NaCl administered as a fast IV bolus dose (within 30 seconds) at 3 or 15 minutes following administration of Esmeron®,
  Other Names: NaCl 0.9%
  Arms: Arm A. Placebo; 3 min after 1 mg/kg Esmeron®; Arm G. Placebo; 15 min after 1 mg/kg Esmeron®; Arm M. Placebo; 3 min after 1.2 mg/kg Esmeron®; Arm S. Placebo; 15 min after 1.2 mg/kg Esmeron®
Drug: Esmeron® — Esmeron® administered at 1 or 1.2 mg/kg as a fast IV bolus (within 10 seconds), dosed according to participant actual body weight.
  Other Names: Zemuron®; Rocuronium bromide

SUMMARY:
The objective of this trial was to explore the dose-response relation of sugammadex (Org 25969; MK-8616) administered for the reversal of neuromuscular blockade (NMB) at 3 and 15 minutes following administration of 1.0 and 1.2 mg/kg of Esmeron® (rocuronium) in participants receiving surgery, classified as American Society of Anesthesiologists (ASA) class 1 (otherwise normal, healthy participant), class 2 (participant with mild systemic disease), or class 3 (participant with a severe systemic disease that limits activity, but is not incapacitating).

DETAILED DESCRIPTION:
In the United States, the highest dose recommended in the package insert of Zemuron® (i.e. the trade name for Esmeron® in the US) is 1.2 mg/kg whereas in Europe it is 1.0 mg/kg. For both doses, dose recommendations for reversal with sugammadex were to be found. Hence, the present trial was set up to explore the dose-response relation of sugammadex given as an NMB reversal agent at 3 and 15 minutes following administration of 1.0 and 1.2 mg/kg of Esmeron® in subjects of ASA 1 to 3. The sub-investigator who performed any subjective safety assessments after anesthesia was to be remained blinded.

ELIGIBILITY:
Inclusion Criteria:

* Participants of ASA class 1 - 3, above or equal to the age of 18 years;
* Participants scheduled for surgical procedures with an anticipated duration of anesthesia of at least 120 minutes, without further need for muscle relaxation other than for intubation;
* Participants scheduled for surgical procedures in supine position;
* Participants who had given written informed consent.

Exclusion Criteria:

* Participants in whom a difficult intubation because of anatomical malformations was expected;
* Participants known or suspected to have neuromuscular disorders impairing neuromuscular blocking and/or significant renal dysfunction;
* Participants known or suspected to have a (family) history of malignant hyperthermia;
* Participants known or suspected to have an allergy to narcotics, muscle relaxants or other medication used during general anesthesia;
* Participants receiving medication known to interfere with neuromuscular blocking agents, such as anticonvulsants and Mg^2+;
* Participants who had already participated in this trial;
* Participants who had participated in another clinical trial, not pre-approved by the Sponsor, within 30 days of entering into this trial;
* Female participants who were pregnant: in females, pregnancy was to be excluded both from medical history and by a human chorionic gonadotropin (hCG) test within 24 hours before surgery except in females who were not of childbearing potential, i.e. at least 2 years menopausal or who had undergone tubal ligation or an hysterectomy;
* Female participants of childbearing potential not using any of the following methods of birth control (for one month): condom or diaphragm with spermicide, vasectomized partner (>6 months), intrauterine device (IUD), abstinence;
* Female participants who were breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2004-03-04 (Actual); Primary Completion 2004-07-20 (Actual); Study Completion 2004-07-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Puhringer FK, Rex C, Sielenkamper AW, Claudius C, Larsen PB, Prins ME, Eikermann M, Khuenl-Brady KS. Reversal of profound, high-dose rocuronium-induced neuromuscular blockade by sugammadex at two different time points: an international, multicenter, randomized, dose-finding, safety assessor-blinded, phase II trial. Anesthesiology. 2008 Aug;109(2):188-97. doi: 10.1097/ALN.0b013e31817f5bc7. PMID 18648227
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/policies-perspectives.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of the N=174 randomized participants, N=173 received treatment. Treated participants are counted as Started in the arm that most accurately describes the treatment received. If no treatment was received (N=1 participant), participants are counted as Started in the arm to which they were randomized.
Pre-assignment Details: N=2 participants (randomized to Arm O) received (rec'd) 8 mg/kg Sugammadex, 3 minutes (min) after 1.2 mg/kg Esmeron® and are counted as Started/Treated in Arm P. Further, N=1 participant (randomized to Arm Q) rec'd 12 mg/kg Sugammadex, 29 min after 1.2 mg/kg Esmeron® and is counted as Started/Treated in Arm W.
Groups:
- Arm G. Placebo; 15 Min After 1 mg/kg Esmeron®: Placebo (single IV bolus) administered 15 min after the bolus intubation dose of 1 mg/kg Esmeron®.
Period: Overall Study
Arm/Group | Arm A. Placebo; 3 Min After 1 mg/kg Esmeron® | Arm B. 2 mg/kg Sugammadex; 3 Min After 1 mg/kg Esmeron® | Arm C. 4 mg/kg Sugammadex; 3 Min After 1 mg/kg Esmeron® | Arm D. 8 mg/kg Sugammadex; 3 Min After 1 mg/kg Esmeron® | Arm E. 12 mg/kg Sugammadex; 3 Min After 1 mg/kg Esmeron® | Arm F. 16 mg/kg Sugammadex; 3 Min After 1 mg/kg Esmeron® | Arm G. Placebo; 15 Min After 1 mg/kg Esmeron® | Arm H. 2 mg/kg Sugammadex; 15 Min After 1 mg/kg Esmeron® | Arm I. 4 mg/kg Sugammadex; 15 Min After 1 mg/kg Esmeron® | Arm J. 8 mg/kg Sugammadex; 15 Min After 1 mg/kg Esmeron® | Arm K. 12 mg/kg Sugammadex; 15 Min After 1 mg/kg Esmeron® | Arm L. 16 mg/kg Sugammadex; 15 Min After 1 mg/kg Esmeron® | Arm M. Placebo; 3 Min After 1.2 mg/kg Esmeron® | Arm N. 2 mg/kg Sugammadex; 3 Min After 1.2 mg/kg Esmeron® | Arm O. 4 mg/kg Sugammadex; 3 Min After 1.2 mg/kg Esmeron® | Arm P. 8 mg/kg Sugammadex; 3 Min After 1.2 mg/kg Esmeron® | Arm Q. 12 mg/kg Sugammadex; 3 Min After 1.2 mg/kg Esmeron® | Arm R. 16 mg/kg Sugammadex; 3 Min After 1.2 mg/kg Esmeron® | Arm S. Placebo; 15 Min After 1.2 mg/kg Esmeron® | Arm T. 2 mg/kg Sugammadex; 15 Min After 1.2 mg/kg Esmeron® | Arm U. 4 mg/kg Sugammadex; 15 Min After 1.2 mg/kg Esmeron® | Arm V. 8 mg/kg Sugammadex; 15 Min After 1.2 mg/kg Esmeron® | Arm W. 12 mg/kg Sugammadex; 15 Min After 1.2 mg/kg Esmeron® | Arm X. 16 mg/kg Sugammadex; 15 Min After 1.2 mg/kg Esmeron®
Started | 5 | 11 | 11 | 11 | 11 | 10 | 3 | 5 | 5 | 5 | 5 | 5 | 5 | 10 | 9 | 13 (N=11 randomized to Arm P. An additional N=2 (randomized to Arm O) are counted as Started in Arm P) | 10 | 11 | 3 | 5 | 5 | 5 | 6 (N=5 randomized to Arm W. An additional N=1 (randomized to Arm Q) is counted as Started in Arm W) | 5
Treated (All participants as treated) | 5 | 11 | 11 | 11 | 11 | 10 | 3 | 5 | 4 | 5 | 5 | 5 | 5 | 10 | 9 | 13 (N=2 (randomized to Arm O) rec'd 8 mg/kg Sugammadex, 3 min after 1.2 mg/kg Esmeron®) | 10 | 11 | 3 | 5 | 5 | 5 | 6 (N=1 (randomized to Arm Q) rec'd 12 mg/kg Sugammadex, 29 min after 1.2 mg/kg Esmeron®) | 5
Completed | 5 | 11 | 11 | 11 | 11 | 10 | 3 | 5 | 4 | 4 | 5 | 5 | 5 | 10 | 9 | 13 | 10 | 11 | 3 | 5 | 5 | 4 | 6 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Includes all participants receiving study treatment. N=2 participants (originally randomized to Arm O), rec'd 8 mg/kg sugammadex, 3 min after 1.2 mg/kg Esmeron® (counted in Arm P). N=1 participant (originally randomized to Arm Q) rec'd 12 mg/kg sugammadex, 29min after 1.2 mg/kg Esmeron® (counted in Arm W).
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A. Placebo; 3 Min After 1 mg/kg Esmeron® | Arm B. 2 mg/kg Sugammadex; 3 Min After 1 mg/kg Esmeron® | Arm C. 4 mg/kg Sugammadex; 3 Min After 1 mg/kg Esmeron® | Arm D. 8 mg/kg Sugammadex; 3 Min After 1 mg/kg Esmeron® | Arm E. 12 mg/kg Sugammadex; 3 Min After 1 mg/kg Esmeron® | Arm F. 16 mg/kg Sugammadex; 3 Min After 1 mg/kg Esmeron® | Arm G. Placebo; 15 Min After 1 mg/kg Esmeron® | Arm H. 2 mg/kg Sugammadex; 15 Min After 1 mg/kg Esmeron® | Arm I. 4 mg/kg Sugammadex; 15 Min After 1 mg/kg Esmeron® | Arm J. 8 mg/kg Sugammadex; 15 Min After 1 mg/kg Esmeron® | Arm K. 12 mg/kg Sugammadex; 15 Min After 1 mg/kg Esmeron® | Arm L. 16 mg/kg Sugammadex; 15 Min After 1 mg/kg Esmeron® | Arm M. Placebo; 3 Min After 1.2 mg/kg Esmeron® | Arm N. 2 mg/kg Sugammadex; 3 Min After 1.2 mg/kg Esmeron® | Arm O. 4 mg/kg Sugammadex; 3 Min After 1.2 mg/kg Esmeron® | Arm P. 8 mg/kg Sugammadex; 3 Min After 1.2 mg/kg Esmeron® | Arm Q. 12 mg/kg Sugammadex; 3 Min After 1.2 mg/kg Esmeron® | Arm R. 16 mg/kg Sugammadex; 3 Min After 1.2 mg/kg Esmeron® | Arm S. Placebo; 15 Min After 1.2 mg/kg Esmeron® | Arm T. 2 mg/kg Sugammadex; 15 Min After 1.2 mg/kg Esmeron® | Arm U. 4 mg/kg Sugammadex; 15 Min After 1.2 mg/kg Esmeron® | Arm V. 8 mg/kg Sugammadex; 15 Min After 1.2 mg/kg Esmeron® | Arm W. 12 mg/kg Sugammadex; 15 Min After 1.2 mg/kg Esmeron® | Arm X. 16 mg/kg Sugammadex; 15 Min After 1.2 mg/kg Esmeron® | Total
Number analyzed (Participants) | 5 | 11 | 11 | 11 | 11 | 10 | 3 | 5 | 4 | 5 | 5 | 5 | 5 | 10 | 9 | 13 | 10 | 11 | 3 | 5 | 5 | 5 | 6 | 5 | 173
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Includes all participants receiving study treatment. N=2 participants (originally randomized to Arm O), rec'd 8 mg/kg sugammadex, 3 min after 1.2 mg/kg Esmeron® (counted in Arm P). N=1 participant (originally randomized to Arm Q) rec'd 12 mg/kg sugammadex, 29min after 1.2 mg/kg Esmeron® (counted in Arm W).
  Years | 49.8 (16.0) | 45.8 (17.9) | 48.4 (16.3) | 46.8 (11.3) | 47.5 (12.8) | 54.9 (17.5) | 43.3 (5.7) | 51.2 (18.9) | 63.0 (6.2) | 45.2 (17.3) | 56.0 (8.9) | 62.4 (7.9) | 57.2 (13.2) | 53.0 (16.2) | 47.9 (21.1) | 52.6 (12.6) | 57.5 (14.6) | 48.7 (15.4) | 48.0 (28.0) | 41.8 (21.3) | 45.0 (17.0) | 44.8 (19.8) | 51.8 (10.3) | 46.0 (22.4) | 50.4 (15.6)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Includes all participants receiving study treatment. N=2 participants (originally randomized to Arm O), rec'd 8 mg/kg sugammadex, 3 min after 1.2 mg/kg Esmeron® (counted in Arm P). N=1 participant (originally randomized to Arm Q) rec'd 12 mg/kg sugammadex, 29min after 1.2 mg/kg Esmeron® (counted in Arm W).
  Participants
    Female | 2 | 3 | 7 | 7 | 5 | 7 | 0 | 2 | 0 | 1 | 1 | 5 | 4 | 6 | 6 | 3 | 4 | 6 | 2 | 1 | 2 | 1 | 1 | 4 | 80
    Male | 3 | 8 | 4 | 4 | 6 | 3 | 3 | 3 | 4 | 4 | 4 | 0 | 1 | 4 | 3 | 10 | 6 | 5 | 1 | 4 | 3 | 4 | 5 | 1 | 93
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Includes all participants receiving study treatment. N=2 participants (originally randomized to Arm O), rec'd 8 mg/kg sugammadex, 3 min after 1.2 mg/kg Esmeron® (counted in Arm P). N=1 participant (originally randomized to Arm Q) rec'd 12 mg/kg sugammadex, 29min after 1.2 mg/kg Esmeron® (counted in Arm W).
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    White | 5 | 11 | 11 | 11 | 10 | 10 | 3 | 5 | 4 | 5 | 5 | 5 | 5 | 10 | 9 | 13 | 10 | 11 | 3 | 5 | 5 | 5 | 5 | 5 | 171
    More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Mean Time From Start of Study Treatment Administration to Recovery of the T4/T1 Ratio to 0.9
Description: Mean time from start of study treatment administration to recovery of participant T4/T1 ratio to 0.9 was assessed through the repeated application (every 15 seconds) of an electrical stimulation protocol. Specifically, 4 electrical stimulations were applied to the ulnar nerve and the magnitude of the twitch response of the adductor pollicis muscle (i.e. thumb twitch response) was assessed. With T4 and T1 referring to the respective magnitude of the fourth and first thumb twitch during nerve stimulation, the T4/T1 ratio indicates the current degree of neuromuscular blockade (NMB) present in the participant as a decimal from 0 (loss of T4 twitch) to 1 (no NMB). Further, reduced recovery time of the T4/T1 ratio to 0.9 indicates faster recovery from NMB. Summary data, originally presented in the format of units "minutes:seconds" (mm:ss), was reformatted to be presented in the single unit of "minutes" (min).
Time Frame: Up to 240 minutes following administration of study treatment
Population: Includes all participants receiving study treatment, having ≥1 post-baseline observation without a major protocol violation. Additionally, N=1 participant was excluded from Arm M due to missing data and N=1 participant was excluded from Arm N due to unreliability of the neuromuscular data.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Arm A. Placebo; 3 Min After 1 mg/kg Esmeron® | Arm B. 2 mg/kg Sugammadex; 3 Min After 1 mg/kg Esmeron® | Arm C. 4 mg/kg Sugammadex; 3 Min After 1 mg/kg Esmeron® | Arm D. 8 mg/kg Sugammadex; 3 Min After 1 mg/kg Esmeron® | Arm E. 12 mg/kg Sugammadex; 3 Min After 1 mg/kg Esmeron® | Arm F. 16 mg/kg Sugammadex; 3 Min After 1 mg/kg Esmeron® | Arm G. Placebo; 15 Min After 1 mg/kg Esmeron® | Arm H. 2 mg/kg Sugammadex; 15 Min After 1 mg/kg Esmeron® | Arm I. 4 mg/kg Sugammadex; 15 Min After 1 mg/kg Esmeron® | Arm J. 8 mg/kg Sugammadex; 15 Min After 1 mg/kg Esmeron® | Arm K. 12 mg/kg Sugammadex; 15 Min After 1 mg/kg Esmeron® | Arm L. 16 mg/kg Sugammadex; 15 Min After 1 mg/kg Esmeron® | Arm M. Placebo; 3 Min After 1.2 mg/kg Esmeron® | Arm N. 2 mg/kg Sugammadex; 3 Min After 1.2 mg/kg Esmeron® | Arm O. 4 mg/kg Sugammadex; 3 Min After 1.2 mg/kg Esmeron® | Arm P. 8 mg/kg Sugammadex; 3 Min After 1.2 mg/kg Esmeron® | Arm Q. 12 mg/kg Sugammadex; 3 Min After 1.2 mg/kg Esmeron® | Arm R. 16 mg/kg Sugammadex; 3 Min After 1.2 mg/kg Esmeron® | Arm S. Placebo; 15 Min After 1.2 mg/kg Esmeron® | Arm T. 2 mg/kg Sugammadex; 15 Min After 1.2 mg/kg Esmeron® | Arm U. 4 mg/kg Sugammadex; 15 Min After 1.2 mg/kg Esmeron® | Arm V. 8 mg/kg Sugammadex; 15 Min After 1.2 mg/kg Esmeron® | Arm W. 12 mg/kg Sugammadex; 15 Min After 1.2 mg/kg Esmeron® | Arm X. 16 mg/kg Sugammadex; 15 Min After 1.2 mg/kg Esmeron®
Number analyzed (Participants) | 5 | 11 | 11 | 11 | 11 | 10 | 3 | 5 | 4 | 5 | 5 | 5 | 4 | 9 | 8 | 11 | 10 | 11 | 3 | 5 | 5 | 5 | 5 | 5
minutes | 108.43 (31.17) | 44.73 (22.18) | 6.93 (2.87) | 2.40 (1.17) | 2.42 (2.12) | 1.77 (1.13) | 127.37 (92.77) | 8.53 (1.12) | 5.47 (3.13) | 1.85 (0.55) | 1.78 (0.87) | 0.93 (0.13) | 122.98 (28.47) | 65.67 (24.58) | 13.78 (7.63) | 3.23 (0.98) | 2.08 (0.85) | 1.32 (0.42) | 139.62 (79.88) | 42.20 (29.33) | 5.97 (2.47) | 2.33 (0.30) | 1.77 (1.18) | 4.73 (6.68)

2. Secondary Outcome: Mean Time From Start of Study Treatment Administration to Recovery of the T4/T1 Ratio to 0.8
Description: Mean time from start of study treatment administration to recovery of participant T4/T1 ratio to 0.8 was assessed through the repeated application (every 15 seconds) of an electrical stimulation protocol. Specifically, 4 electrical stimulations were applied to the ulnar nerve and the magnitude of the twitch response of the adductor pollicis muscle (i.e. thumb twitch response) was assessed. With T4 and T1 referring to the respective magnitude of the fourth and first thumb twitch during nerve stimulation, the T4/T1 ratio indicates the current degree of NMB present in the participant as a decimal from 0 (loss of T4 twitch) to 1 (no NMB). Further, reduced recovery time of the T4/T1 ratio to 0.8 indicates faster recovery from NMB. Summary data, originally presented in the format of units "minutes:seconds" (mm:ss), was reformatted to be presented in the single unit of "minutes" (min).
Time Frame: Up to 200 minutes following administration of study treatment
Population: Includes all participants receiving study treatment, having ≥1 post-baseline observation without a major protocol violation.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Arm A. Placebo; 3 Min After 1 mg/kg Esmeron® | Arm B. 2 mg/kg Sugammadex; 3 Min After 1 mg/kg Esmeron® | Arm C. 4 mg/kg Sugammadex; 3 Min After 1 mg/kg Esmeron® | Arm D. 8 mg/kg Sugammadex; 3 Min After 1 mg/kg Esmeron® | Arm E. 12 mg/kg Sugammadex; 3 Min After 1 mg/kg Esmeron® | Arm F. 16 mg/kg Sugammadex; 3 Min After 1 mg/kg Esmeron® | Arm G. Placebo; 15 Min After 1 mg/kg Esmeron® | Arm H. 2 mg/kg Sugammadex; 15 Min After 1 mg/kg Esmeron® | Arm I. 4 mg/kg Sugammadex; 15 Min After 1 mg/kg Esmeron® | Arm J. 8 mg/kg Sugammadex; 15 Min After 1 mg/kg Esmeron® | Arm K. 12 mg/kg Sugammadex; 15 Min After 1 mg/kg Esmeron® | Arm L. 16 mg/kg Sugammadex; 15 Min After 1 mg/kg Esmeron® | Arm M. Placebo; 3 Min After 1.2 mg/kg Esmeron® | Arm N. 2 mg/kg Sugammadex; 3 Min After 1.2 mg/kg Esmeron® | Arm O. 4 mg/kg Sugammadex; 3 Min After 1.2 mg/kg Esmeron® | Arm P. 8 mg/kg Sugammadex; 3 Min After 1.2 mg/kg Esmeron® | Arm Q. 12 mg/kg Sugammadex; 3 Min After 1.2 mg/kg Esmeron® | Arm R. 16 mg/kg Sugammadex; 3 Min After 1.2 mg/kg Esmeron® | Arm S. Placebo; 15 Min After 1.2 mg/kg Esmeron® | Arm T. 2 mg/kg Sugammadex; 15 Min After 1.2 mg/kg Esmeron® | Arm U. 4 mg/kg Sugammadex; 15 Min After 1.2 mg/kg Esmeron® | Arm V. 8 mg/kg Sugammadex; 15 Min After 1.2 mg/kg Esmeron® | Arm W. 12 mg/kg Sugammadex; 15 Min After 1.2 mg/kg Esmeron® | Arm X. 16 mg/kg Sugammadex; 15 Min After 1.2 mg/kg Esmeron®
Number analyzed (Participants) | 5 | 11 | 11 | 11 | 11 | 10 | 3 | 5 | 4 | 5 | 5 | 5 | 5 | 10 | 8 | 11 | 10 | 11 | 3 | 5 | 5 | 5 | 5 | 5
minutes | 98.23 (28.82) | 40.00 (20.47) | 5.90 (2.40) | 1.87 (0.73) | 1.57 (1.35) | 1.43 (0.97) | 91.53 (43.73) | 6.23 (1.23) | 4.10 (2.60) | 1.45 (0.43) | 1.33 (0.50) | 0.93 (0.13) | 129.85 (39.48) | 60.85 (21.13) | 8.52 (2.80) | 2.80 (1.02) | 1.73 (0.82) | 1.20 (0.27) | 121.03 (63.07) | 33.95 (23.02) | 4.42 (1.38) | 1.98 (0.27) | 1.72 (1.07) | 1.27 (0.60)

3. Secondary Outcome: Mean Time From Start of Study Treatment Administration to Recovery of the T4/T1 Ratio to 0.7
Description: Mean time from start of study treatment administration to recovery of participant T4/T1 ratio to 0.7 was assessed through the repeated application (every 15 seconds) of an electrical stimulation protocol. Specifically, 4 electrical stimulations were applied to the ulnar nerve and the magnitude of the twitch response of the adductor pollicis muscle (i.e. thumb twitch response) was assessed. With T4 and T1 referring to the respective magnitude of the fourth and first thumb twitch during nerve stimulation, the T4/T1 ratio indicates the current degree of NMB present in the participant as a decimal from 0 (loss of T4 twitch) to 1 (no NMB). Further, reduced recovery time of the T4/T1 ratio to 0.7 indicates faster recovery from NMB. Summary data, originally presented in the format of units "minutes:seconds" (mm:ss), was reformatted to be presented in the single unit of "minutes" (min).
Time Frame: Up to 180 minutes following administration of study treatment
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Arm A. Placebo; 3 Min After 1 mg/kg Esmeron® | Arm B. 2 mg/kg Sugammadex; 3 Min After 1 mg/kg Esmeron® | Arm C. 4 mg/kg Sugammadex; 3 Min After 1 mg/kg Esmeron® | Arm D. 8 mg/kg Sugammadex; 3 Min After 1 mg/kg Esmeron® | Arm E. 12 mg/kg Sugammadex; 3 Min After 1 mg/kg Esmeron® | Arm F. 16 mg/kg Sugammadex; 3 Min After 1 mg/kg Esmeron® | Arm G. Placebo; 15 Min After 1 mg/kg Esmeron® | Arm H. 2 mg/kg Sugammadex; 15 Min After 1 mg/kg Esmeron® | Arm I. 4 mg/kg Sugammadex; 15 Min After 1 mg/kg Esmeron® | Arm J. 8 mg/kg Sugammadex; 15 Min After 1 mg/kg Esmeron® | Arm K. 12 mg/kg Sugammadex; 15 Min After 1 mg/kg Esmeron® | Arm L. 16 mg/kg Sugammadex; 15 Min After 1 mg/kg Esmeron® | Arm M. Placebo; 3 Min After 1.2 mg/kg Esmeron® | Arm N. 2 mg/kg Sugammadex; 3 Min After 1.2 mg/kg Esmeron® | Arm O. 4 mg/kg Sugammadex; 3 Min After 1.2 mg/kg Esmeron® | Arm P. 8 mg/kg Sugammadex; 3 Min After 1.2 mg/kg Esmeron® | Arm Q. 12 mg/kg Sugammadex; 3 Min After 1.2 mg/kg Esmeron® | Arm R. 16 mg/kg Sugammadex; 3 Min After 1.2 mg/kg Esmeron® | Arm S. Placebo; 15 Min After 1.2 mg/kg Esmeron® | Arm T. 2 mg/kg Sugammadex; 15 Min After 1.2 mg/kg Esmeron® | Arm U. 4 mg/kg Sugammadex; 15 Min After 1.2 mg/kg Esmeron® | Arm V. 8 mg/kg Sugammadex; 15 Min After 1.2 mg/kg Esmeron® | Arm W. 12 mg/kg Sugammadex; 15 Min After 1.2 mg/kg Esmeron® | Arm X. 16 mg/kg Sugammadex; 15 Min After 1.2 mg/kg Esmeron®
Number analyzed (Participants) | 5 | 11 | 11 | 11 | 11 | 10 | 3 | 5 | 4 | 5 | 5 | 5 | 5 | 10 | 8 | 11 | 10 | 11 | 3 | 5 | 5 | 5 | 5 | 5
minutes | 91.58 (27.43) | 36.43 (17.22) | 4.55 (1.43) | 1.58 (0.70) | 1.13 (0.12) | 1.27 (0.52) | 81.70 (34.18) | 5.28 (0.77) | 3.28 (1.62) | 1.25 (0.15) | 1.28 (0.42) | 0.93 (0.13) | 122.90 (36.23) | 54.43 (17.33) | 7.45 (2.82) | 2.42 (0.85) | 1.62 (0.80) | 1.18 (0.22) | 111.37 (53.03) | 24.15 (13.00) | 3.08 (0.90) | 1.58 (0.35) | 1.67 (0.97) | 1.22 (0.57)

4. Secondary Outcome: Number of Participants Experiencing an Adverse Event
Description: The number of participants experiencing an adverse event (AE) was assessed. An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of an investigational product, whether or not considered related to the investigational product.
Time Frame: Up to 7 days following administration of study treatment
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A. Placebo; 3 Min After 1 mg/kg Esmeron® | Arm B. 2 mg/kg Sugammadex; 3 Min After 1 mg/kg Esmeron® | Arm C. 4 mg/kg Sugammadex; 3 Min After 1 mg/kg Esmeron® | Arm D. 8 mg/kg Sugammadex; 3 Min After 1 mg/kg Esmeron® | Arm E. 12 mg/kg Sugammadex; 3 Min After 1 mg/kg Esmeron® | Arm F. 16 mg/kg Sugammadex; 3 Min After 1 mg/kg Esmeron® | Arm G. Placebo; 15 Min After 1 mg/kg Esmeron® | Arm H. 2 mg/kg Sugammadex; 15 Min After 1 mg/kg Esmeron® | Arm I. 4 mg/kg Sugammadex; 15 Min After 1 mg/kg Esmeron® | Arm J. 8 mg/kg Sugammadex; 15 Min After 1 mg/kg Esmeron® | Arm K. 12 mg/kg Sugammadex; 15 Min After 1 mg/kg Esmeron® | Arm L. 16 mg/kg Sugammadex; 15 Min After 1 mg/kg Esmeron® | Arm M. Placebo; 3 Min After 1.2 mg/kg Esmeron® | Arm N. 2 mg/kg Sugammadex; 3 Min After 1.2 mg/kg Esmeron® | Arm O. 4 mg/kg Sugammadex; 3 Min After 1.2 mg/kg Esmeron® | Arm P. 8 mg/kg Sugammadex; 3 Min After 1.2 mg/kg Esmeron® | Arm Q. 12 mg/kg Sugammadex; 3 Min After 1.2 mg/kg Esmeron® | Arm R. 16 mg/kg Sugammadex; 3 Min After 1.2 mg/kg Esmeron® | Arm S. Placebo; 15 Min After 1.2 mg/kg Esmeron® | Arm T. 2 mg/kg Sugammadex; 15 Min After 1.2 mg/kg Esmeron® | Arm U. 4 mg/kg Sugammadex; 15 Min After 1.2 mg/kg Esmeron® | Arm V. 8 mg/kg Sugammadex; 15 Min After 1.2 mg/kg Esmeron® | Arm W. 12 mg/kg Sugammadex; 15 Min After 1.2 mg/kg Esmeron® | Arm X. 16 mg/kg Sugammadex; 15 Min After 1.2 mg/kg Esmeron®
Number analyzed (Participants) | 5 | 11 | 11 | 11 | 11 | 10 | 3 | 5 | 4 | 5 | 5 | 5 | 5 | 10 | 9 | 13 | 10 | 11 | 3 | 5 | 5 | 5 | 6 | 5
Participants | 5 | 5 | 7 | 7 | 8 | 7 | 2 | 4 | 3 | 4 | 3 | 4 | 3 | 5 | 7 | 5 | 6 | 9 | 3 | 2 | 4 | 1 | 3 | 3

ADVERSE EVENTS:
Time Frame: Up to 7 days following administration of study treatment
Description: Includes all participants receiving study treatment. N=2 participants (originally randomized to Arm O), rec'd 8 mg/kg sugammadex, 3 min after 1.2 mg/kg Esmeron® (counted in Arm P). N=1 participant (originally randomized to Arm Q) rec'd 12 mg/kg sugammadex, 29min after 1.2 mg/kg Esmeron® (counted in Arm W).
Groups:
- Arm A. Placebo; 3 Min After 1 mg/kg Esmeron: Placebo (single IV bolus) administered 3 min after the bolus intubation dose of 1 mg/kg Esmeron®.
- Arm B. 2 mg/kg Sugammadex; 3 Min After 1 mg/kg Esmeron: Sugammadex (2 mg/kg; single IV bolus) administered 3 min after the bolus intubation dose of 1 mg/kg Esmeron®.
- Arm C. 4 mg/kg Sugammadex; 3 Min After 1 mg/kg Esmeron: Sugammadex (4 mg/kg; single IV bolus) administered 3 min after the bolus intubation dose of 1 mg/kg Esmeron®.
- Arm D. 8 mg/kg Sugammadex; 3 Min After 1 mg/kg Esmeron: Sugammadex (8 mg/kg; single IV bolus) administered 3 min after the bolus intubation dose of 1 mg/kg Esmeron®.
- Arm E. 12 mg/kg Sugammadex; 3 Min After 1 mg/kg Esmeron: Sugammadex (12 mg/kg; single IV bolus) administered 3 min after the bolus intubation dose of 1 mg/kg Esmeron®.
- Arm F. 16 mg/kg Sugammadex; 3 Min After 1 mg/kg Esmeron: Sugammadex (16 mg/kg; single IV bolus) administered 3 min after the bolus intubation dose of 1 mg/kg Esmeron®.
- Arm G. Placebo; 15 Min After 1 mg/kg Esmeron: Placebo (single IV bolus) administered 15 min after the bolus intubation dose of 1 mg/kg Esmeron®.
- Arm H. 2 mg/kg Sugammadex; 15 Min After 1 mg/kg Esmeron: Sugammadex (2 mg/kg; single IV bolus) administered 15 min after the bolus intubation dose of 1 mg/kg Esmeron®.
- Arm I. 4 mg/kg Sugammadex; 15 Min After 1 mg/kg Esmeron: Sugammadex (4 mg/kg; single IV bolus) administered 15 min after the bolus intubation dose of 1 mg/kg Esmeron®.
- Arm J. 8 mg/kg Sugammadex; 15 Min After 1 mg/kg Esmeron: Sugammadex (8 mg/kg; single IV bolus) administered 15 min after the bolus intubation dose of 1 mg/kg Esmeron®.
- Arm K. 12 mg/kg Sugammadex; 15 Min After 1 mg/kg Esmeron: Sugammadex (12 mg/kg; single IV bolus) administered 15 min after the bolus intubation dose of 1 mg/kg Esmeron®.
- Arm L. 16 mg/kg Sugammadex; 15 Min After 1 mg/kg Esmeron: Sugammadex (16 mg/kg; single IV bolus) administered 15 min after the bolus intubation dose of 1 mg/kg Esmeron®.
- Arm M. Placebo; 3 Min After 1.2 mg/kg Esmeron: Placebo (single IV bolus) administered 3 min after the bolus intubation dose of 1.2 mg/kg Esmeron®.
- Arm N. 2 mg/kg Sugammadex; 3 Min After 1.2 mg/kg Esmeron: Sugammadex (2 mg/kg; single IV bolus) administered 3 min after the bolus intubation dose of 1.2 mg/kg Esmeron®.
- Arm O. 4 mg/kg Sugammadex; 3 Min After 1.2 mg/kg Esmeron: Sugammadex (4 mg/kg; single IV bolus) administered 3 min after the bolus intubation dose of 1.2 mg/kg Esmeron®.
- Arm P. 8 mg/kg Sugammadex; 3 Min After 1.2 mg/kg Esmeron: Sugammadex (8 mg/kg; single IV bolus) administered 3 min after the bolus intubation dose of 1.2 mg/kg Esmeron®.
- Arm Q. 12 mg/kg Sugammadex; 3 Min After 1.2 mg/kg Esmeron: Sugammadex (12 mg/kg; single IV bolus) administered 3 min after the bolus intubation dose of 1.2 mg/kg Esmeron®.
- Arm R. 16 mg/kg Sugammadex; 3 Min After 1.2 mg/kg Esmeron: Sugammadex (16 mg/kg; single IV bolus) administered 3 min after the bolus intubation dose of 1.2 mg/kg Esmeron®.
- Arm S. Placebo; 15 Min After 1.2 mg/kg Esmeron: Placebo (single IV bolus) administered 15 min after the bolus intubation dose of 1.2 mg/kg Esmeron®.
- Arm T. 2 mg/kg Sugammadex; 15 Min After 1.2 mg/kg Esmeron: Sugammadex (2 mg/kg; single IV bolus) administered 15 min after the bolus intubation dose of 1.2 mg/kg Esmeron®.
- Arm U. 4 mg/kg Sugammadex; 15 Min After 1.2 mg/kg Esmeron: Sugammadex (4 mg/kg; single IV bolus) administered 15 min after the bolus intubation dose of 1.2 mg/kg Esmeron®.
- Arm V. 8 mg/kg Sugammadex; 15 Min After 1.2 mg/kg Esmeron: Sugammadex (8 mg/kg; single IV bolus) administered 15 min after the bolus intubation dose of 1.2 mg/kg Esmeron®.
- Arm W. 12 mg/kg Sugammadex; 15 Min After 1.2 mg/kg Esmeron: Sugammadex (12 mg/kg; single IV bolus) administered 15 min after the bolus intubation dose of 1.2 mg/kg Esmeron®.
- Arm X. 16 mg/kg Sugammadex; 15 Min After 1.2 mg/kg Esmeron: Sugammadex (16 mg/kg; single IV bolus) administered 15 min after the bolus intubation dose of 1.2 mg/kg Esmeron®.
Arm/Group | Arm A. Placebo; 3 Min After 1 mg/kg Esmeron | Arm B. 2 mg/kg Sugammadex; 3 Min After 1 mg/kg Esmeron | Arm C. 4 mg/kg Sugammadex; 3 Min After 1 mg/kg Esmeron | Arm D. 8 mg/kg Sugammadex; 3 Min After 1 mg/kg Esmeron | Arm E. 12 mg/kg Sugammadex; 3 Min After 1 mg/kg Esmeron | Arm F. 16 mg/kg Sugammadex; 3 Min After 1 mg/kg Esmeron | Arm G. Placebo; 15 Min After 1 mg/kg Esmeron | Arm H. 2 mg/kg Sugammadex; 15 Min After 1 mg/kg Esmeron | Arm I. 4 mg/kg Sugammadex; 15 Min After 1 mg/kg Esmeron | Arm J. 8 mg/kg Sugammadex; 15 Min After 1 mg/kg Esmeron | Arm K. 12 mg/kg Sugammadex; 15 Min After 1 mg/kg Esmeron | Arm L. 16 mg/kg Sugammadex; 15 Min After 1 mg/kg Esmeron | Arm M. Placebo; 3 Min After 1.2 mg/kg Esmeron | Arm N. 2 mg/kg Sugammadex; 3 Min After 1.2 mg/kg Esmeron | Arm O. 4 mg/kg Sugammadex; 3 Min After 1.2 mg/kg Esmeron | Arm P. 8 mg/kg Sugammadex; 3 Min After 1.2 mg/kg Esmeron | Arm Q. 12 mg/kg Sugammadex; 3 Min After 1.2 mg/kg Esmeron | Arm R. 16 mg/kg Sugammadex; 3 Min After 1.2 mg/kg Esmeron | Arm S. Placebo; 15 Min After 1.2 mg/kg Esmeron | Arm T. 2 mg/kg Sugammadex; 15 Min After 1.2 mg/kg Esmeron | Arm U. 4 mg/kg Sugammadex; 15 Min After 1.2 mg/kg Esmeron | Arm V. 8 mg/kg Sugammadex; 15 Min After 1.2 mg/kg Esmeron | Arm W. 12 mg/kg Sugammadex; 15 Min After 1.2 mg/kg Esmeron | Arm X. 16 mg/kg Sugammadex; 15 Min After 1.2 mg/kg Esmeron
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/11 | 0/11 | 0/11 | 0/11 | 0/10 | 0/3 | 0/5 | 0/4 | 0/5 | 0/5 | 0/5 | 0/5 | 0/10 | 0/9 | 0/13 | 0/10 | 0/11 | 0/3 | 0/5 | 0/5 | 0/5 | 0/6 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 1/11 | 0/11 | 1/11 | 0/11 | 3/10 | 0/3 | 0/5 | 0/4 | 0/5 | 0/5 | 1/5 | 1/5 | 0/10 | 2/9 | 0/13 | 1/10 | 1/11 | 0/3 | 0/5 | 1/5 | 0/5 | 0/6 | 0/5
Other Adverse Events (participants affected / at risk) | 5/5 | 5/11 | 7/11 | 7/11 | 8/11 | 6/10 | 2/3 | 4/5 | 3/4 | 4/5 | 3/5 | 4/5 | 3/5 | 5/10 | 7/9 | 5/13 | 6/10 | 9/11 | 3/3 | 2/5 | 3/5 | 1/5 | 3/6 | 3/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A. Placebo; 3 Min After 1 mg/kg Esmeron (N=5) | Arm B. 2 mg/kg Sugammadex; 3 Min After 1 mg/kg Esmeron (N=11) | Arm C. 4 mg/kg Sugammadex; 3 Min After 1 mg/kg Esmeron (N=11) | Arm D. 8 mg/kg Sugammadex; 3 Min After 1 mg/kg Esmeron (N=11) | Arm E. 12 mg/kg Sugammadex; 3 Min After 1 mg/kg Esmeron (N=11) | Arm F. 16 mg/kg Sugammadex; 3 Min After 1 mg/kg Esmeron (N=10) | Arm G. Placebo; 15 Min After 1 mg/kg Esmeron (N=3) | Arm H. 2 mg/kg Sugammadex; 15 Min After 1 mg/kg Esmeron (N=5) | Arm I. 4 mg/kg Sugammadex; 15 Min After 1 mg/kg Esmeron (N=4) | Arm J. 8 mg/kg Sugammadex; 15 Min After 1 mg/kg Esmeron (N=5) | Arm K. 12 mg/kg Sugammadex; 15 Min After 1 mg/kg Esmeron (N=5) | Arm L. 16 mg/kg Sugammadex; 15 Min After 1 mg/kg Esmeron (N=5) | Arm M. Placebo; 3 Min After 1.2 mg/kg Esmeron (N=5) | Arm N. 2 mg/kg Sugammadex; 3 Min After 1.2 mg/kg Esmeron (N=10) | Arm O. 4 mg/kg Sugammadex; 3 Min After 1.2 mg/kg Esmeron (N=9) | Arm P. 8 mg/kg Sugammadex; 3 Min After 1.2 mg/kg Esmeron (N=13) | Arm Q. 12 mg/kg Sugammadex; 3 Min After 1.2 mg/kg Esmeron (N=10) | Arm R. 16 mg/kg Sugammadex; 3 Min After 1.2 mg/kg Esmeron (N=11) | Arm S. Placebo; 15 Min After 1.2 mg/kg Esmeron (N=3) | Arm T. 2 mg/kg Sugammadex; 15 Min After 1.2 mg/kg Esmeron (N=5) | Arm U. 4 mg/kg Sugammadex; 15 Min After 1.2 mg/kg Esmeron (N=5) | Arm V. 8 mg/kg Sugammadex; 15 Min After 1.2 mg/kg Esmeron (N=5) | Arm W. 12 mg/kg Sugammadex; 15 Min After 1.2 mg/kg Esmeron (N=6) | Arm X. 16 mg/kg Sugammadex; 15 Min After 1.2 mg/kg Esmeron (N=5)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A. Placebo; 3 Min After 1 mg/kg Esmeron (N=5) | Arm B. 2 mg/kg Sugammadex; 3 Min After 1 mg/kg Esmeron (N=11) | Arm C. 4 mg/kg Sugammadex; 3 Min After 1 mg/kg Esmeron (N=11) | Arm D. 8 mg/kg Sugammadex; 3 Min After 1 mg/kg Esmeron (N=11) | Arm E. 12 mg/kg Sugammadex; 3 Min After 1 mg/kg Esmeron (N=11) | Arm F. 16 mg/kg Sugammadex; 3 Min After 1 mg/kg Esmeron (N=10) | Arm G. Placebo; 15 Min After 1 mg/kg Esmeron (N=3) | Arm H. 2 mg/kg Sugammadex; 15 Min After 1 mg/kg Esmeron (N=5) | Arm I. 4 mg/kg Sugammadex; 15 Min After 1 mg/kg Esmeron (N=4) | Arm J. 8 mg/kg Sugammadex; 15 Min After 1 mg/kg Esmeron (N=5) | Arm K. 12 mg/kg Sugammadex; 15 Min After 1 mg/kg Esmeron (N=5) | Arm L. 16 mg/kg Sugammadex; 15 Min After 1 mg/kg Esmeron (N=5) | Arm M. Placebo; 3 Min After 1.2 mg/kg Esmeron (N=5) | Arm N. 2 mg/kg Sugammadex; 3 Min After 1.2 mg/kg Esmeron (N=10) | Arm O. 4 mg/kg Sugammadex; 3 Min After 1.2 mg/kg Esmeron (N=9) | Arm P. 8 mg/kg Sugammadex; 3 Min After 1.2 mg/kg Esmeron (N=13) | Arm Q. 12 mg/kg Sugammadex; 3 Min After 1.2 mg/kg Esmeron (N=10) | Arm R. 16 mg/kg Sugammadex; 3 Min After 1.2 mg/kg Esmeron (N=11) | Arm S. Placebo; 15 Min After 1.2 mg/kg Esmeron (N=3) | Arm T. 2 mg/kg Sugammadex; 15 Min After 1.2 mg/kg Esmeron (N=5) | Arm U. 4 mg/kg Sugammadex; 15 Min After 1.2 mg/kg Esmeron (N=5) | Arm V. 8 mg/kg Sugammadex; 15 Min After 1.2 mg/kg Esmeron (N=5) | Arm W. 12 mg/kg Sugammadex; 15 Min After 1.2 mg/kg Esmeron (N=6) | Arm X. 16 mg/kg Sugammadex; 15 Min After 1.2 mg/kg Esmeron (N=5)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye irritation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (3) | 2 (2) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 4 (4) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 3 (4) | 2 (2) | 4 (4) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Airway complication of anaesthesia (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaesthetic complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 2 (4) | 4 (4) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (2) | 2 (3) | 2 (3) | 5 (7) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Delayed recovery from anaesthesia (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periorbital haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural hypertension (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural hypotension (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Heart rate decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Red blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Restlessness (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oliguria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor recognizes the right of the investigators to publish, but all publications must be based on data validated and released by the Sponsor. Any such scientific paper, presentation, or other communication concerning the clinical trial described in this protocol will first be submitted to the Sponsor, at least six weeks ahead of estimated publication or presentation, for written consent, which shall not be withheld unreasonably.